CLINICAL TRIAL: NCT05659628
Title: Phase Ib Clinical Study of CD19 CAR-T Expressing IL-7 and CCL19 Combined With Tislelizumab in the Treatment of Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: CD19 CAR-T Expressing IL-7 and CCL19 Combined With Anti-PD1 in RR-DLBCL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ningbo101
Record Dates: First submitted 2022-11-26; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T combined with anti-PD1 treatment group (Experimental): CD19-7×19 CAR-T combined with Tislelizumab
  Interventions: Combination Product: CD19-7×19 CAR-T combined with Tislelizumab

INTERVENTIONS:
Combination Product: CD19-7×19 CAR-T combined with Tislelizumab — Participants will receive 2×106/Kg CD19-7×19 CAR-T cells infusion and Tislelizumab 200mg every 21 days for 6 cycle on the 31st day after CAR-T infusion.

SUMMARY:
The goal of this clinical trial is to test CD19-7×19 CAR-T cells combined with Tislelizumab in refractory and relapsed diffuse large B lymphoma. The main question[s] it aims to answer are:

question 1：What is the safety of CD19-7×19 CAR-T cells combined with Tislelizumab in the treatment of relapsed or refractory diffuse large B-cell lymphoma.

question 2：What is the efficacy of CD19-7×19 CAR-T cells combined with Tislelizumab in the treatment of relapsed or refractory diffuse large B-cell lymphoma.

Participants will be asked to receive clinical evaluation before CAR-T, including physical examination, blood routine test, biochemical test, imaging test, etc.Peripheral blood lymphocytes will be collected for preparation of CAR-T cells after enrollment. Pretreatment chemotherapy with fludarabine and cyclophosphamide will be used before CAR-T infusion. On the 31st day after CAR-T infusion, Tislelizumab 200mg was given once every 21 days for 6 cycles. Participants will be required to report concomitant medication and adverse events, and their disease was evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, upper limit 75, male or female;
2. ECOG score 0-3;
3. Histologically confirmed diffuse large B-cell lymphoma (DLBCL) [diagnostic criteria according to WHO 2008];
4. CD19 positive (immunohistochemistry or flow cytometry).
5. DLBCL refractory or relapse is defined as: complete remission is not achieved after 2-line treatment; let What disease progress occurs during treatment, or the disease stability time is equal to or less than 6 months; Or autologous hematopoietic stem Disease progression or recurrence within 12 months after cell transplantation;
6. Previous treatment for patients with diffuse large B cell lymphoma must include rituximab (CD20 monoclonal antibody) and anthracyclines;
7. At least one measurable lesion is required, and any lymph node lesion with a length greater than 1.5cm or extranodal lesion is required If any length diameter is greater than 1.0 cm, the lesions on PET-CT scan have uptake (SUV is larger than liver blood pool);
8. Absolute value of peripheral blood neutrophils ≥ 1000/ μ l. Platelets ≥ 45000/ μ l
9. Heart, liver and kidney functions: creatinine < 1.5mg/dL; ALT/AST Less than 2.5 times of normal upper limit; Total bilirubin < 1.5mg/dL; Cardiac ejection fraction (EF) ≥ 50%;
10. Have sufficient understanding and voluntarily sign the informed consent form;
11. People with fertility must be willing to use contraceptive methods;
12. According to the judgment of the researcher, the expected survival period is at least 4 months;
13. Willing to follow the visit schedule, administration plan, laboratory inspection and other test steps.

Exclusion Criteria:

1. Have a history of other tumors;
2. Autologous hematopoietic stem cell transplantation was performed within 6 weeks;
3. Any target CAR-T treatment was performed within 3 months before this CAR-T treatment;
4. Previously used any commercially available PD-1 monoclonal antibody;
5. Cytotoxic drugs, glucocorticoids and other targeted drugs were received within 2 weeks before cell collection;
6. Active autoimmune diseases;
7. Uncontrollable active bacterial and fungal infections;
8. HIV infection and syphilis infection; Active hepatitis B or hepatitis C: hepatitis B: HBV-DNA ≥ 1000 IU/mL; Hepatitis C: HCV RNA is positive and liver function is abnormal.
9. Known central nervous system lymphoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events profile | Measured from start of treatment until 28 days after last dose.
  Number of participants with adverse events. Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 will be tabulated.
Objective Response Rate | up to 3 months
  Proportion of CR and PR subjects will be assessed at 3 months post-infusion.

SECONDARY OUTCOMES:
Progress free survival time | up to 24 months
  To measure the duration of response over a follow-up period of 24 months.
Overall survival | up to 24 months
  OS will be assessed from the first chimeric antigen receptor T cells (CAR-T) given to death or last follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Zhejiang University, Ningbo First Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No